CLINICAL TRIAL: NCT05457400
Title: A Randomized, Double-blind, Active-controlled, Cross-over Study to Assess the Effect of the Sugar Substitute "ENSO 16" on Glucose Metabolism Parameters in Healthy Subjects
Brief Title: ENSO 16 - Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alpha Republic GmbH (Industry)
Collaborators: Vienna General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 00070007
Record Dates: First submitted 2022-03-21; First posted 2022-07-14 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Sugar; Blood, Low
Keywords: Sugar Substitutes; Fibers; Blood Glucose Rise; Blood Glucose Level; Polyols; Blood Glucose Spike
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Intervention Model Description: The objective of this study is to evaluate differences in glucose metabolism parameters after oral administration of 30g glucose or 30g ENSO16. Blood samples will be be collected from 15 male or female subjects at defined time points (0 - 15 - 30 - 45 - 60 - 90 - 120
  - 180 minutes; 3 min at each time point). Individual plasma glucose, insulin and C-peptide concentrations are going to be evaluated and statistically assessed. Subjects will also be asked to complete a questionnaire regarding their digestion after oral intake of ENSO 16 or glucose defined timepoints.
Who Masked: Investigator
Masking Description: The study medication will be provided in identical looking bottles. Because of the completely identical appearance and smell (white, powdery substance and sweet smell), no difference can be perceived by the investigators or subjects. The bottles will be labelled with the respective labels as shown in chapter 8.1.6. Unblinding will be performed after the database lock (e.g. all pseudonymized data for statistical analysis entered into an Excel and/or SPSS sheet). Emergency envelopes will be provided from the sponsor to the Department of Clinical Pharmacology if emergency unblinding is necessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENSO 16 (Active Comparator): The participants receive 30g ENSO 16 dissolved in 200 mL water and blood will be collected at defined time points (0 - 15 - 30 - 45 - 60 - 90 - 120 - 180 minutes; ±3 min at each time point).
  Interventions: Drug: ENSO 16
- Glucose Powder (Active Comparator): The participants receive Glucose in the same dosage and blood is also taken at the same time points.
  Interventions: Drug: Glucose Powder

INTERVENTIONS:
Drug: ENSO 16 — 30 g ENSO 16 dissolved in Water
  Arms: ENSO 16
Drug: Glucose Powder — 30 g Glucose Powder dissolved in Water
  Arms: Glucose Powder

SUMMARY:
The objective of this study is to evaluate differences in glucose metabolism parameters after oral administration of 30g glucose or 30g ENSO16. Blood samples will be be collected from 15 male or female subjects at defined time points (0 - 15 - 30 - 45 - 60 - 90 - 120

- 180 minutes; 3 min at each time point). Individual plasma glucose, insulin and C-peptide concentrations are going to be evaluated and statistically assessed. Subjects will also be asked to complete a questionnaire regarding their digestion after oral intake of ENSO 16 or glucose defined timepoints.

DETAILED DESCRIPTION:
This is a randomized, double-blind, active-controlled, cross-over study to assess the effect of the sugar substitute "ENSO 16" on glucose metabolism parameters in healthy male or female subjects. 15 healthy subects ≥ 18 years will be included and 30 g of ENSO 16 or 30 g glucose will be orally administered to assess the impact on markers of glucose metabolism. The study medication will be dissolved in 200 mL tap water. After randomization, subjects will receive ENSO 16 (group A) or glucose (group B) on the first study day. Following a wash-out period of at least on week, subjects will receive glucose (group A) or ENSO 16 (group B) on the second study day. A screening examination (inclusion/ exclusion criteria, medical history, etc.) will be done on the first study day before the study medication will be administered. The study medication will be administered after an overnight fast of at least 10h. Subjects will receive a venular cannula and blood is going to be collected at 8 pre-defined timepoints (0 - 15 - 30 - 45 - 60 - 90 - 120 - 180 minutes; 3 min at each time point). In total, 192 mL of blood are going to be collected per study participant. Study participants will also have to fill in a questionnaire to rate gastrointestinal symptoms using a checklist including the following questions: ((a) abdominal pain, (b) nausea, (c) vomiting, (d) diarrhoea, (e) abdominal rumbling, (f) bloating, (g) belching and (h) flatulence. Participants were asked to choose between "no symptom" (0 points), "mild symptoms" (1 point) and "severe symptoms" (2 points) for each question at each time point.

Primary Endpoint To test the effect of orally administered ENSO 16 (30 g) or glucose (30 g) on plasma glucose levels. The area under the curve (AUC) of plasma glucose profiles (0-60 min) will be compared between different study days.

Null and alternative hypotheses:

H0: There is no difference in blood glucose AUC (0-60 min) between glucose and ENSO 16. H1: There is a difference in blood glucose AUC (0-60 min) between glucose and ENSO 16. Sample size calculation No formal sample size calculation could be performed for this trial as ENSO 16 has never been tested on glucose metabolism parameters in a clinical trial. There is evidence that sugar substitutes have to be studied separately because sweeteners differ considerably in their chemical structure and their physiologic effect on glucose metabolism. However, based on a cross-over trial with the sugar substitute xylitol at high doses, a sample size of 12 was appropriate to detect significant differences in outcome parameters. Based on these study results and on available statistical recommendations, a sample size of 15 was chosen, which is considered to be appropriate for this cross over trial to detect significant differences in the main outcome parameters if present. Statistical methodology Calculation of the AUC (0-60 min) for plasma glucose, insulin and Cpeptide profiles. Paired T-tests or Wilcoxon signed rank tests (for skewed distributions) will be applied to describe differences between treatments (glucose and ENSO 16)

ELIGIBILITY:
Inclusion Criteria:

* Ability of subject to understand the character and individual consequences of the study;
* Signed informed consent before the start of any specific study procedures;
* Age ≥18 years;
* BMI 18-25 and healthy
* Fasting blood glucose ≤ 100mg/dL (point of care device)

Exclusion Criteria:

* Substance or alcohol abuse
* Smoking
* Regular intake of medication (except oral contraceptives) including over the counter drugs within 2 weeks before study day 1
* Chronic medical illness
* Food allergies and dietary restrictions
* Pregnancy
* Participation in another clinical trial 3 weeks before study day 1

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Effect on blood sugar | 2 weeks
  To test the effect of orally administered ENSO 16 (30 g) or glucose (30 g) on plasma glucose levels. The area under the curve (AUC) of plasma glucose profiles (0-60 min) will be compared between different study days.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik für Klinische Pharmakologie,, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Depends on the resources of the sponsor organization
Supporting Information: CSR

REFERENCES:
- [Derived] Lutnik M, Weisshaar S, Mussbacher LM, Steiner D, Wolzt M. The substitute ENSO 16 has low impact on glucose metabolism in healthy humans: a randomized, double-blind, active-controlled, cross-over trial. Sci Rep. 2024 Jun 24;14(1):14534. doi: 10.1038/s41598-024-65560-w. PMID 38914694